CLINICAL TRIAL: NCT07082075
Title: Joint Hyperlaxity and Volar Plate Dynamics: MRI-Based Comparative Evaluation of the PIP Joint
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, Professor, Hacettepe University
Other Study IDs: KA22/286
Record Dates: First submitted 2025-05-28; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Hypermobility, Joint
Keywords: volar plate; hypermobility; biomechanics
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The volar plate (VP) is a key stabilizer of the proximal interphalangeal joint (PIPJ), and its biomechanical behavior may be altered in individuals with joint hypermobility.

Objective: This study aimed to evaluate the spatial dynamics of the VP and its relationship with the center of joint motion and flexor digitorum profundus (FDP) tendon in individuals with and without joint hyperlaxity using MRI.

Methods: Thirty-two healthy volunteers (16 hyperlax, 16 controls) underwent MRI imaging of both index fingers at five flexion angles (0°, 30°, 60°, 90°, full flexion) and under passive and isometric loading conditions. Key parameters measured included distances from the joint center to VP attachments, VP-FDP tendon distance, and the length between VP ends.

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years

Exclusion Criteria:

* any history of acute or overuse injuries to the examined hand,
* any prior surgical procedures on the examined upper extremity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and hypermobility volunteers
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The Distance Between the Center of Motion (CoM) and the VPLip and VPTip | baseline
  The distances between the center of motion (CoM) and the volar lip of the middle phalanx base (VPLip), and between the CoM and the proximal end of the volar plate at its attachment to the volar base of the proximal phalanx (VPTip), were measured using RadiAnt DICOM Viewer software (version 2024.1) in various PIPJ angles.
The Distance Between VPLip and VPTip | baseline
  The distance between the volar lip of the middle phalanx base (VPLip), and the proximal end of the volar plate at its attachment to the volar base of the proximal phalanx (VPTip) measured using RadiAnt DICOM Viewer software (version 2024.1) in various PIPJ angles. The purpose of this measurement was to observe how the distance between the two ends of the volar plate changes with varying joint angles.
The Distance Between Volar Plate (VP) and FDP Tendon | baseline
  The distance between the midpoint of the volar plate (VP) and the flexor digitorum profundus (FDP) tendon was measured using RadiAnt DICOM Viewer software (version 2024.1) at various proximal interphalangeal joint (PIPJ) angles. The purpose of this measurement was to observe how this distance changes across different flexion angles.
Changes Observed During Grasping and Isometric Contraction | baseline
  Measurements at all flexion angles were conducted under two conditions: while passively grasping a cylindrical object (without force) and during isometric contraction (with force).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can not be ethical.